CLINICAL TRIAL: NCT06945822
Title: Characterizing the Host Response to Leptospirosis for Better Diagnosis and Prognosis - NIHFI
Acronym: NIHFI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre Terrritorial Hospitalier Gaston Bourret (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-077; 2024-A02827-40 (Other: ID-RCB)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Leptospirosis
Keywords: biomarkers; New Caledonia; infection
MeSH Terms: conditions — Leptospirosis; Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals coming to the emergency department of the CHT (Other): Individuals coming to the emergency department of the Centre Hospitalier Territorial de New Caledonia:
  * Either with suspected leptospirosis with signs and symptoms
  * Or healthy and coming for a traumatology and orthopedics consultation, and showing no infectious signs.
  Interventions: Other: Blood sample; Other: Urine Sample

INTERVENTIONS:
Other: Blood sample — For febrile patients with confirmed (group 1) or refuted (group 2) diagnosis of leptospirosis:
  - At D0, D1, D3 and D15 a 20-ml blood sample
  For healthy patients (group 3):
  - At D0 and D15: a 20-ml blood sample
Other: Urine Sample — For all participants, a 5-ml urine sample at D0

SUMMARY:
Leptospirosis is a zoonosis found worldwide, but particularly in humid subtropical and tropical zones. It is caused by pathogenic bacteria of the Leptospira species of the spirochete family. It is estimated that there are over a million cases of leptospirosis worldwide each year, with 60,000 deaths. These figures place leptospirosis among the most dangerous bacterial zoonoses in the world.

The disease affects the most disadvantaged populations, and also inflicts its burden on domestic and farm animals. To this day, however, leptospirosis remains a neglected disease, poorly understood because it has been little studied.

Human leptospirosis initially presents as a febrile syndrome, with fever, headache, myalgia and joint pain. These symptoms are very similar to those observed in influenza, dengue fever and other acute febrile illnesses, making diagnosis very difficult.

Delayed initiation of antibiotic therapy, a treatment recommended by the WHO, is associated with the development of severe forms of leptospirosis. Indeed, in 10% of cases, leptospirosis evolves into severe forms, which are still poorly described, but which result in haemorrhage, multivisceral failure (lungs, kidneys, liver) and a drastic increase in the case-fatality rate. In 2023, 152 cases of leptospirosis were reported in New Caledonia. Of these, 130 people (85%) were hospitalized and 4 deaths were recorded (2.6%).

For patients suffering from leptospirosis, it is therefore important to be able to make the diagnosis quickly, ideally as soon as symptoms appear. It is also crucial to be able to monitor, or even prevent, the development of severe forms of the disease, to ensure optimal patient care.

DETAILED DESCRIPTION:
The goal of this study is to identify diagnostic and prognostic biomarkers based on host response to human leptospirosis in New Caledonia. To achieve this goal, Individuals coming to the emergency department of the Centre Hospitalier Territorial de Nouvelle-Calédonie will be recruited either with suspected leptospirosis with signs and symptoms or healthy showing no infectious signs.

For febrile patients with confirmed (group 1) or refuted (group 2) diagnosis of leptospirosis:

* At D0: a 20-ml blood sample and a 5-ml urine sample
* At D1, D3 and D15: a 20-ml blood sample

For healthy patients (group 3):

* At D0: a 20-ml blood sample and a 5-ml urine sample
* At D15: a 20-ml blood sample.

The analyses to be carried out are :

* Host-pathogen sequencing,
* Metagenomics,
* Transcriptomics,
* Metabolomics,
* And cytokine assays to study the host immune response.

ELIGIBILITY:
Inclusion Criteria:

For all participants :

* Be able to consent,
* Have received information and given written consent,
* Be covered by a social security plan. For groups 1 & 2: febrile individuals
* Have suspected leptospirosis associated with fever (axillary temperature over 38°C) and a clinical picture of suspected leptospirosis (myalgia, headache...). After inclusion, febrile participants will be divided into 2 groups when the diagnosis of leptospirosis is confirmed. The 2 groups are defined as follows:

Group 1: leptospirosis

- Individual with leptospirosis confirmed by PCR, MAT, or isolation (2013 Center For Disease Control and Prevention (CDC) laboratory criteria for a confirmed diagnosis).

Group 2: MFA, with absence of leptospirosis

All individuals in Group 2 will have tests as part of their MFA diagnosis, depending on their symptomatology:

* Other acute bacterial zoonotic infection: Infection confirmed by paired serology or double PCR (2 targets).
* Acute arboviral infection: dengue, chikungunya or Zika virus confirmed by CDC Trioplex PCR in a patient with consistent serology or positive 2nd target PCR.
* Acute respiratory viral infection: Viral agent confirmed by MFA multiplex PCR. For group 3: healthy individuals
* Apyretic individuals, no symptoms of infection or inflammatory disease in the last 28 days.

Exclusion Criteria:

individuals :

* with a chronic inflammatory disease,
* undergoing concomitant antibiotic and/or anti-inflammatory treatment, or under medical care incompatible with the purpose of the study,
* pregnant or breast-feeding women,
* persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care and persons admitted to a health or social institution,
* Adults subject to a legal protection measure or unable to express their consent
* Persons not affiliated to a social security scheme or beneficiaries of such a scheme
* Hospitalized for more than 48 hours,
* Hospitalized or operated on in the previous 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Identify diagnostic and prognostic biomarkers based on host response to human leptospirosis in New Caledonia. | 4 years
  transcriptome study by sequencing host mRNA at different times, in the blood and urine of individuals suspected of having leptospirosis
Identify diagnostic and prognostic biomarkers based on host response to human leptospirosis in New Caledonia. | 4 years
  level of cytokines present at different times, in the blood and urine of individuals suspected of having leptospirosis
Identify diagnostic and prognostic biomarkers based on host response to human leptospirosis in New Caledonia. | 4 years
  identification of the Leptospira spp. serogroup by sequencing bacterial DNA or PCR at different times, in the blood and urine of individuals suspected of having leptospirosis

SECONDARY OUTCOMES:
Develop and validate biomarkers that have already been identified for accurate diagnosis of leptospirosis of varying clinical severity. | 4 years
  Transcriptome study using host mRNA sequencing
Develop and validate biomarkers that have already been identified for accurate diagnosis of leptospirosis of varying clinical severity. | 4 years
  Level of cytokines or other markers previously identified as biomarkers of severity.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Veyrier, PhD, Study Director — Institut Pasteur de Nouvelle-Calédonie; Cécile Cazorla, MD, Principal Investigator — Centre Hospitalier Territorial Gaston-Bourret